CLINICAL TRIAL: NCT03632577
Title: High Flow Oxygen (HFO) VERSUS Non Invasive Ventilation (NIV) Associated to Automated Flow Oxygen Titration (AFOT) After Extubation in Patient With Respiratory Risk: Non-inferiority Prospective Comparative Study
Brief Title: High Flow Oxygen VERSUS Non Invasive Ventilation Associated to Automated Flow Oxygen Titration After Patient Extubation
Acronym: RespiFLOW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC31/16/8769
Record Dates: First submitted 2018-03-25; First posted 2018-08-15 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Respiratory Disease
Keywords: High Flow Oxygen; Non Invasive Ventilation; Automated Flow Oxygen Titration; respiratory risk
MeSH Terms: conditions — Respiration Disorders | interventions — Noninvasive Ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Flow Oxygen (HFO) (Experimental): HFO is a mix tap of air and oxygen. It permits to control FiO2 and generated controlled high flow air until 60/min. Air and oxygen are mixed, warmed, humidified and issued to patient by a warming monopod inspiratory circuit to nasal cannulas of a large diameter. Expiration is free.
  Interventions: Device: High Flow Oxygen (HFO)
- Non Invasive Ventilation (NIV) (Active Comparator): NIV was already evaluated in post-extubation. This technic is now used in daily consolidation processing after extubation because it provides a ventilator help with two levels of pressure helping in respiratory work. Adding Automated Flow Oxygen Titration could optimized patient's oxygenation and reduce workload of caregivers
  Interventions: Device: Non Invasive Ventilation (NIV)

INTERVENTIONS:
Device: High Flow Oxygen (HFO) — HFO is a mix tap of air and oxygen. It permits to control FiO2 and generated controlled high flow air until 60/min. Air and oxygen are mixed, warmed, humidified and issued to patient by a warming monopod inspiratory circuit to nasal cannulas of a large diameter. Expiration is free.
  Arms: High Flow Oxygen (HFO)
Device: Non Invasive Ventilation (NIV) — NIV was already evaluated in post-extubation. This technic is now used in daily consolidation processing after extubation because it provides a ventilator help with two levels of pressure helping in respiratory work. Adding Automated Flow Oxygen Titration could optimized patient's oxygenation and reduce workload of caregivers.
  Arms: Non Invasive Ventilation (NIV)

SUMMARY:
Extubation stay at high risk of reintubation even scheduled and in the best condition of hematosis. Re-intubation's rate in main studies in chronic obstructive diseases reach to 20% and it is associated to a higher mortality, higher pneumonia under mechanic ventilation, and higher duration of hospitalization especially in intensive care units.

Place of NIV in this situation is still on evaluation. A recent meta-analysis demonstrates that use of NIV in post-extubation in COPD seems to decrease re-intubation rate.

HFO, thanks to its properties (oxygen, humidification and heat with high flow) could be useful in this population in ventilatory weaning. Compared to oxygen conventional therapy with high-concentration mask, HFO seems to be as efficient and better tolerated. A recent study shows that HFO is non-inferior to NVI in post-extubation in patient with high risk of re-intubation.

Furthermore, oxygenation in post-extubation should be optimized to avoid hypoxemia and hypercapnia in this patient at risk of hypoventilation. Place of AFOT could improve hematosis by providing adapted flow of oxygen to each patient.

The investigator choose the hypothesis for this study that HFO is as effective and tolerated in post-extubation than NIV with AFOT.

DETAILED DESCRIPTION:
A recent meta-analysis demonstrates that use of NIV in post-extubation in obstructive chronic bronchopathies seems to decrease re-intubation rate.

High Flow Oxygen, thanks to its properties (oxygen, humidification and heat with high flow) could be useful in this population in ventilatory weaning. Compared to oxygen conventional therapy with high-concentration mask, High Flow Oxygen seems to be as efficient and better tolerated . A recent study shows that High Flow Oxygen is non-inferior to Non Invasive Ventilation in post-extubation in patient with high risk of re-intubation.

Furthermore, oxygenation in post-extubation should be optimized to avoid hypoxemia and hypercapnia in this patient at risk of hypoventilation.

ELIGIBILITY:
Inclusion Criteria:

* Patient with respiratory disease suspected or proved (COPD, asthma, bronchiectasis, cystic fibrosis, interstitial pneumonia, obstructive insufficient respiratory, restrictive insufficient respiratory) when an extubation is scheduled.
* Patient who signed the informed consent
* Patient affiliated to social insurance

Exclusion Criteria:

* Pregnant woman
* Terminal extubation
* NIV at home before intubation (non-exclusion of continue positive airway pressure: CPAP)
* Tracheotomy
* Patient under trusteeship, guardianship or safeguard of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-10-15 (Actual)

PRIMARY OUTCOMES:
Primary outcome: Tolerance of each dispositive | Hours 0
  Comfort scale (from 0 to 100 : 0 is totally uncomfortable - 100 : comfortable)
Primary outcome: Tolerance of each dispositive | Hours 6
  Comfort scale (from 0 to 100 : 0 is totally uncomfortable - 100 : comfortable)
Primary outcome: Tolerance of each dispositive | Hours 24
  Comfort scale (from 0 to 100 : 0 is totally uncomfortable - 100 : comfortable)
Primary outcome: Tolerance of each dispositive | Hours 48
  Comfort scale (from 0 to 100 : 0 is totally uncomfortable - 100 : comfortable)

SECONDARY OUTCOMES:
Dyspnea scale of Borg | Hours 6
  Dyspnea score which is a quantitative measure of the perception of effort during a physical exercise. The measure is a rating on a scale from 0 to 10 attached to different words of appreciation: "very light, difficult, painful ..." effort. This global measurement, based on the physical and psychological sensations of the person, takes into account the physical condition, the environmental conditions and the level of general fatigue. The scale between 0 and 10 was designed to approximate the heart rate of a healthy young adult (effort 8 represents 80% of the CF).
Dyspnea scale of Borg | Hours 24
  Dyspnea score which is a quantitative measure of the perception of effort during a physical exercise. The measure is a rating on a scale from 0 to 10 attached to different words of appreciation: "very light, difficult, painful ..." effort. This global measurement, based on the physical and psychological sensations of the person, takes into account the physical condition, the environmental conditions and the level of general fatigue. The scale between 0 and 10 was designed to approximate the heart rate of a healthy young adult (effort 8 represents 80% of the CF).
Dyspnea scale of Borg | Hours 48
  Dyspnea score which is a quantitative measure of the perception of effort during a physical exercise. The measure is a rating on a scale from 0 to 10 attached to different words of appreciation: "very light, difficult, painful ..." effort. This global measurement, based on the physical and psychological sensations of the person, takes into account the physical condition, the environmental conditions and the level of general fatigue. The scale between 0 and 10 was designed to approximate the heart rate of a healthy young adult (effort 8 represents 80% of the CF).
Treatment's failure defined as use of NVI in HFO group or use of HFO in NVI group | Month 3
  defined by reintubation or exchange of treatment or premature discontinuation of treatment
Hematosis : PaO2, PaCO2, pH | hours 6
  Measurement of PaO2, PaCO2 and pH
Hematosis : PaO2, PaCO2, pH | hours 24
  Measurement of PaO2, PaCO2 and pH
Hematosis : PaO2, PaCO2, pH | hours 48
  Measurement of PaO2, PaCO2 and pH
Duration of hospitalization in intensive care units, reanimation, hospital after extubation. | Month 3
  Measurement of hospitalization in intensive care units in days
Mortality in ICU (continuous monitoring unit) | Month 3
  Measurement of mortality
Mortality in hospital | Month 3
  Measurement of mortality
Mortality at M1 and M3 | Month 1
  Measurement of mortality
Mortality at M1 and M3 | Month 3
  Measurement of mortality
Use of another technic (HFO or NVI) in time | hours 72
  Duration of use of the device (VNI, OHD) at H72
Respiratory congestion (number of fibroscopy for airway's desobstruction, number of respiratory kinesitherapy consults, radiological atelectasis) | month 3
  Measurement of respiratory congestion by : number of fibroscopy for airway's desobstruction, number of respiratory kinesitherapy consults and radiological atelectasis
New intubation rate at H48 | Hours 48
  New intubation rate at H48
New intubation rate at H72 | Hours 72
  New intubation rate at H72
SpO2 stability | hours 48
  Percentage of time spent below 88% and above 92% of SpO2
SpO2 stability | hours 72
  Percentage of time spent below 88% and above 92% of SpO2

CONTACTS AND LOCATIONS:
Overall Officials: Elise Noel-Savina, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Larrey, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bajaj A, Rathor P, Sehgal V, Shetty A. Efficacy of noninvasive ventilation after planned extubation: A systematic review and meta-analysis of randomized controlled trials. Heart Lung. 2015 Mar-Apr;44(2):150-7. doi: 10.1016/j.hrtlng.2014.12.002. Epub 2015 Jan 13. PMID 25592206
- [Background] Tiruvoipati R, Lewis D, Haji K, Botha J. High-flow nasal oxygen vs high-flow face mask: a randomized crossover trial in extubated patients. J Crit Care. 2010 Sep;25(3):463-8. doi: 10.1016/j.jcrc.2009.06.050. Epub 2009 Sep 24. PMID 19781896
- [Background] Brotfain E, Zlotnik A, Schwartz A, Frenkel A, Koyfman L, Gruenbaum SE, Klein M. Comparison of the effectiveness of high flow nasal oxygen cannula vs. standard non-rebreather oxygen face mask in post-extubation intensive care unit patients. Isr Med Assoc J. 2014 Nov;16(11):718-22. PMID 25558703
- [Background] Frat JP, Thille AW, Mercat A, Girault C, Ragot S, Perbet S, Prat G, Boulain T, Morawiec E, Cottereau A, Devaquet J, Nseir S, Razazi K, Mira JP, Argaud L, Chakarian JC, Ricard JD, Wittebole X, Chevalier S, Herbland A, Fartoukh M, Constantin JM, Tonnelier JM, Pierrot M, Mathonnet A, Beduneau G, Deletage-Metreau C, Richard JC, Brochard L, Robert R; FLORALI Study Group; REVA Network. High-flow oxygen through nasal cannula in acute hypoxemic respiratory failure. N Engl J Med. 2015 Jun 4;372(23):2185-96. doi: 10.1056/NEJMoa1503326. Epub 2015 May 17. PMID 25981908
- [Background] Hernandez G, Vaquero C, Colinas L, Cuena R, Gonzalez P, Canabal A, Sanchez S, Rodriguez ML, Villasclaras A, Fernandez R. Effect of Postextubation High-Flow Nasal Cannula vs Noninvasive Ventilation on Reintubation and Postextubation Respiratory Failure in High-Risk Patients: A Randomized Clinical Trial. JAMA. 2016 Oct 18;316(15):1565-1574. doi: 10.1001/jama.2016.14194. PMID 27706464